CLINICAL TRIAL: NCT06051448
Title: Harnessing Resilience in Adults With Primary Mitochondrial Disease: A Pilot Study Investigating the Feasibility of the Promoting Resilience in Stress Management (PRISM) and Clinical-focused Narrative (CFN) Interventions
Brief Title: Promoting Resilience in Stress Management (PRISM) and Clinical-focused Narrative (CFN) Pilot in Adults With Primary Mitochondrial Disease (PMD).
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: North American Mitochondrial Disease Consortium (NAMDC) (Unknown); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-020222; U54NS078059-12 (NIH)
Record Dates: First submitted 2023-09-12; First posted 2023-09-25 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial Encephalomyopathies; MELAS; MERRF
MeSH Terms: conditions — Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial Encephalomyopathies; MELAS Syndrome; MERRF Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promoting Resilience in Stress Management (PRISM) (Active Comparator)
  Interventions: Behavioral: Promoting Resilience in Stress Management (PRISM)
- Clinical-focused narrative (CFN) (Active Comparator)
  Interventions: Behavioral: Clinical-focused narrative (CFN)

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management (PRISM) — This program teaches the four pillars of resilience (stress management, goal setting, cognitive restructuring, and benefit-finding) in a one-on-one training program consisting of four 20-30 minute sessions occurring once weekly.
  Arms: Promoting Resilience in Stress Management (PRISM)
Behavioral: Clinical-focused narrative (CFN) — This program consists of questions posed to adults with primary mitochondrial disease at regular mitochondrial medicine center visits. Specific topics will be discussed at each session. This consists four 20-30 minute sessions occurring once weekly.
  Arms: Clinical-focused narrative (CFN)

SUMMARY:
The goal of this study is to find the best way to help people with primary mitochondrial disease deal with the stress of their condition, and to help these people be better able to "bounce back," or be resilient. In order to do this, the investigators are going to test two interventions (an intervention means that it aims to change something): Promoting Resilience in Stress Management (PRISM) and clinical-focused narrative (CFN) intervention.

DETAILED DESCRIPTION:
The investigators are going to test two interventions in this pilot study. The first is called Promoting Resilience in Stress Management (PRISM). The second is called clinical-focused narrative (CFN) intervention. These interventions involve talking with the researcher about several specific topics.

Participants will join six virtual study visits. They will be assigned to the PRISM group or the CFN group. During the first study visit, participants will learn about the study and will fill out consent forms if they want to participate. In the next four visits, participants will receive one of the study interventions (PRISM or CFN). Some interventions will be supported with a digital app for participants to track progress and review what was talked about in the intervention. The sixth virtual study visit will be a discussion group that happens a couple months after participants finish the intervention.

Participants will also be sent several surveys to complete. One set of surveys is sent just once after the participant enrolls in the study. Another set of surveys is sent after the participant enrolls and again after the participant finishes the interventions.

The study team will review participants' medical records to confirm they have primary mitochondrial disease and to review the genetic diagnosis. If participants do not have copies of their own medical records or if the study team does not already have access to them, the study team will ask participants to sign a release form to obtain a copy of the medical records and/or genetic testing report.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18 years old
2. Capable of giving consent, or there is a legally authorized representative capable of giving consent on the subject behalf and if appropriate, assent.
3. Able to speak and read English
4. Able to participate in Web- and App-based interventions
5. Confirmed molecular diagnosis of primary mitochondrial disease

Exclusion Criteria:

1. Suspected but no molecular diagnosis primary mitochondrial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Determine mean score on validated scale assessing resilience in those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The Connor-Davidson Resilience Scale (CD-RISC) is a validated measure to assess resilience. Possible scores range from 0-100 (higher scores reflecting greater resilience). Mean scores will be calculated on scales administered to subjects before the intervention and scales administered after intervention completion.
Determine change in mean in scores on validated scale assessing resilience between those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The Connor-Davidson Resilience Scale (CD-RISC) is a validated measure to assess resilience. Possible scores range from 0-100 (higher scores reflecting greater resilience). Mean scores calculated on scales administered before the intervention will be compared to mean scores on scales administered after completion of the intervention.
Determine variability in scores on validated scale assessing resilience between those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The Connor-Davidson Resilience Scale (CD-RISC) is a validated measure to assess resilience. Possible scores range from 0-100 (higher scores reflecting greater resilience). Variability in scores of scales collected before starting and after completion of the interventions will be calculated.
Determine mean scores on validated scale assessing coping in those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The Family Crisis Oriented Personal Scale (F-COPES) is a validated measure to assess coping. Possible scores range from 30 to 150 (higher scores reflect higher levels of coping and problem-solving ability). Mean scores will be calculated on scales administered to subjects before the intervention and scales administered after intervention completion.
Determine change in mean scores on validated scale assessing coping between those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The Family Crisis Oriented Personal Scale (F-COPES) is a validated measure to assess coping. Possible scores range from 30 to 150 (higher scores reflect higher levels of coping and problem-solving ability). Mean scores calculated on scales administered before the intervention will be compared to mean scores on scales administered after completion of the intervention.
Determine variability in scores on a validated scale assessing coping between those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The Family Crisis Oriented Personal Scale (F-COPES) is a validated measure to assess coping. Possible scores range from 30 to 150 (higher scores reflect higher levels of coping and problem-solving ability). Variability in scores of scales collected before starting and after completion of the interventions will be calculated.
Determine mean scores on validated scale assessing quality of life in those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The 36-Item Short Form Survey Instrument (SF-36) is a validated measure to assess quality of life. Possible scores range from 0-100 (higher scores reflect a more favorable health state). Mean scores calculated on scales administered before the intervention will be compared to mean scores on scales administered after completion of the intervention.
Determine change in mean in scores on validated scale assessing quality of life between those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The 36-Item Short Form Survey Instrument (SF-36) is a validated measure to assess quality of life. Possible scores range from 0-100 (higher scores reflect a more favorable health state). Mean scores will be calculated on scales administered to subjects before the intervention and scales administered after intervention completion.
Determine variability in scores on a validated scale assessing quality of life between those who receive PRISM and those who receive CFN. | Up to 3 months after the first intervention
  The 36-Item Short Form Survey Instrument (SF-36) is a validated measure to assess quality of life. Possible scores range from 0-100 (higher scores reflect a more favorable health state). Variability in scores of scales collected before starting and after completion of the interventions will be calculated.

SECONDARY OUTCOMES:
Explore participant experience with PRISM and CFN and assess their acceptability among adults with primary mitochondrial disease. | Three months after completing the intervention, discussion groups will occur.
  Semi-structured interviews will be conducted at discussion groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M McCormick, MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study, without direct patient identifiers will be released to an NIH data repository for the purpose of facilitating data sharing according to NIH policy
Time Frame: By the time of publication
Access Criteria: Anonymized participant data will be released to an NIH repository and will be available upon request.